CLINICAL TRIAL: NCT05866328
Title: Online Training Program on Social Cognition for Patients With Schizophrenia
Brief Title: Online TP (Training Program) on SC (Social Cognition) for Schizophrenia
Acronym: TP;SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Collaborators: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Francisco Pulido, Professor of Psychiatry, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ULaguna
Record Dates: First submitted 2019-09-11; First posted 2023-05-19 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Social Cognition
Keywords: rehabilitation; schizophrenia; emotional adjustment; theory of mind
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training; Palliative Care; Myo-Inositol-1-Phosphate Synthase

STUDY DESIGN:
Intervention Model Description: Cognitive rehabilitation with a cognitive training program
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Experimental: ET and IPS Control: IPS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Experimental Group (e-Motional Training and Individual Placement and Support)
  Interventions: Other: Cognitive Rehabilitation and Individual Placement and Support
- Control (No Intervention): Control Group (Individual Placement and Support)

INTERVENTIONS:
Other: Cognitive Rehabilitation and Individual Placement and Support — Cognitive Rehabilitation and Individual Placement and Support
  Other Names: CR and IPS
  Arms: Intervention

SUMMARY:
Randomized controlled trial. Sixty-five participants (83% with schizophrenia or bipolar disorder) were recruited from community mental health teams. Fifty-seven met criteria and agreed to participate in the study. The conditions of cognitive rehabilitation were assigned randomly with support employment CR + IPS (n = 28) and IPS alone (n = 29). Cogpack program was used. Two groups were followed at 8 and 12 months after the baseline.

DETAILED DESCRIPTION:
This work was developed in the island of Tenerife (Spain) within a public service specialised in labour integration of people with disabilities in which an IPS team was set up in 2005. The study was carried out in collaboration with the units of community mental health of the island. These units carry out the control of people with serious mental illnesses including pharmacological treatment and psychosocial programming. All research procedures were approved by the Medicine Committee of Canary Health Services.

The follow-up period for the data collection was set between 2013 and 2014. Employment specialists belong to a public institution specialized in work disability.Sixty-five participants but only 57 signed written informed consent and completed the baseline. Two groups were assigned randomly:one with support employment and cognitive rehabilitation the second group with IPS alone

ELIGIBILITY:
Inclusion Criteria:

Participants had to:

1. comply with the state definitions of severe mental illness (SMI), which includes an ICD-10 (World Health Organization, 1992) diagnosis of F20- 29 (schizophrenia, schizotypal, delusional and other non-mood psychotic disorders) and F31-F32.3 (major mood affective disorders)
2. have previous difficulties to maintain a job
3. currently want a competitive job and
4. accept the job search starts

Exclusion Criteria:

People with no Severe mental illness and not want to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Ekman 60 Faces Test total score changes | At baseline and after 1 year treatment
  Minimum 0 and maximum 60. Between 20-40 years average 51.43, cut-off point 45, below deficit. Between 40-60 years, average 51.20, cut-off point 43, below deficit.
Hinting Task total score changes | At baseline and after 1 year treatment
  Total 1 minimum 0 and maximum 20. Total 2 minimum 0 and maximum 10. Cut-off point 18, less deficit.
Happé Strange Stories Test total score changes | At baseline and after 1 year treatment
  Total control minimum 0 and maximum 16. Total theory of mind minimum 0 and maximum 16. Cut-off point 14, below the deficit.
Faux Pas Recognition Test total score changes | At baseline and after 1 year treatment
  FP stories and C questions, C stories and FP questions and C stories and C questions minimum 0 and maximum 20. FP stories and FP questions minimum 0 and maximum 60. Cut-off point without errors 54 and with errors 48, lower deficit scores.
Ambiguous Intentions and Hostility Questionnaire total score changes | At baseline and after 1 year treatment
  Hostility, anger, guilt and aggression minimum 1 and maximum 5. Intentionality minimum 1 and maximum 6. Calculate the mean.
Movie for the Assessment of Social Cognition total score changes | At baseline and after 1 year treatment
  Minimum 0 and maximum 42.
Screening for Cognitive Impairment in Psychiatry (SCIP-S) total score changes | At baseline and after 1 year treatment
  Minimum 1 and maximum 99, very low range 1-2.5 and low range 2.5-15. The deterioration depends on the scale.
Positive and Negative Symptom Scale (PANSS) total score changes | At baseline and after 1 year treatment
  Positive and negative subscales minimum 7 and maximum 49. General psychopathology subscale minimum 16 and maximum 112. Composite subscale minimum -42 and maximum +42. Categorize subtype positive >0 and negative <0.

SECONDARY OUTCOMES:
Employment | Up to 12 months in 2021
  Number of jobs

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Rodriguez Pulido, PHD MD, Study Director — University of La Laguna
Locations (1):
- Francisco Rodriguez Pulido, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publicate the results in a International Journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2019-2020
Access Criteria: International Journal

REFERENCES:
- [Result] Vazquez-Campo M, Marono Y, Lahera G, Mateos R, Garcia-Caballero A. e-Motional Training(R): Pilot study on a novel online training program on social cognition for patients with schizophrenia. Schizophr Res Cogn. 2016 Mar 12;4:10-17. doi: 10.1016/j.scog.2015.11.007. eCollection 2016 Jun. PMID 28740808
- [Result] Marono Souto Y, Vazquez Campo M, Diaz Llenderrozas F, Rodriguez Alvarez M, Mateos R, Garcia Caballero A. Randomized Clinical Trial with e-MotionalTraining(R) 1.0 for Social Cognition Rehabilitation in Schizophrenia. Front Psychiatry. 2018 Feb 26;9:40. doi: 10.3389/fpsyt.2018.00040. eCollection 2018. PMID 29535646
- [Derived] Rodriguez Pulido F, Caballero Estebaranz N, Garcia Caballero AA, Gonzalez Davila E, Leon Palacin C, Hernandez Alvarez de Sotomayor MDC, Lopez Reig S, Vilchez de Leon PI. Social cognition and emotional rehabilitation in participants with schizofrenia. Front Psychiatry. 2023 Nov 8;14:1250933. doi: 10.3389/fpsyt.2023.1250933. eCollection 2023. PMID 38025483

DOCUMENTS (3):
  • Study Protocol (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT05866328/Prot_003.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT05866328/SAP_001.pdf
  • Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT05866328/ICF_002.pdf